CLINICAL TRIAL: NCT05170568
Title: A Phase I Open-label, Dose-escalation Trial of PA3-17 Injection in Adult Patients With CD7-positive Relapsed/Refractory Lymphoid Hematologic Malignancies
Brief Title: PA3-17 Injection Treatment of Adult Patients With CD7-positive Relapsed/Refractory Lymphoid Hematologic Malignancies
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: PersonGen BioTherapeutics (Suzhou) Co., Ltd. (Industry)
Collaborators: The First Affiliated Hospital of Zhengzhou University (Other); Peking University People's Hospital (Other); Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other); Hematology Hospital of Chinese Academy of Medical Sciences (Hematology Research Center of Chinese Academy of Medical Sciences) (Unknown); Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PG-CART-07-001 (1)
Record Dates: First submitted 2021-12-24; First posted 2021-12-28 (Actual); Last update posted 2022-11-01 (Actual); Status verified 2022-10

CONDITIONS: CD7-positive Relapsed/Refractory Lymphoid Hematologic Malignancies

STUDY DESIGN:
Intervention Model Description: PA3-17 injection
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- T cell injection targeting CD7 chimeric antigen receptor (Experimental)
  Interventions: Biological: T cell injection targeting CD7 chimeric antigen receptor

INTERVENTIONS:
Biological: T cell injection targeting CD7 chimeric antigen receptor — The subjects, who sign the informed consent forms and been screened by inclusion/exclusion criteria, will be assigned into 0.5 × 106, 2.0 × 106 and 4.0 × 106 CAR-T/kg groups in order of sequence. And the subjects will be administered once.
  Other Names: PA3-17 injection

SUMMARY:
This is a Phase I, open-label, dose-escalation clinical study with the primary objective of evaluating the safety and tolerability of PA3-17 injection in adult subjects with CD7-positive relapsed/refractory lymphoid hematologic malignancies. The secondary objectives are as follows: to evaluate the proliferation and in vivo persistence of CD7-targeted chimeric antigen receptor T (CAR-T) cells after injection of PA3-17; to evaluate the proportion of CD7-positive cells in peripheral blood after injection of PA3-17; to preliminarily evaluate the efficacy of PA3-17 injection in adult subjects with CD7-positive relapsed/refractory lymphoid hematologic malignancies; to evaluate the immunogenicity of PA3-17 injection; and to explore the applicable dose in Phase II trial.

DETAILED DESCRIPTION:
Approximately 5 sites are planned to be selected for the clinical trial. The subjects, who sign the informed consent forms and been screened by inclusion/exclusion criteria, will be assigned into 0.5 × 10^6, 2.0 × 10^6 and 4.0 × 10^6 CAR-T/kg groups in order of sequence. And the subjects will be administered once. Dose escalation will follow 3 + 3 design and 3-6 subjects in each group will complete a single dose. Within the same dose group, the next subject will be administered after the previous subject has completed at least 14 days of safety observation. After the last subject in each dose group has completed the dose-limiting toxicity (DLT) assessment window of 28 days after single dose, the enrollment and treatment for the next dose group may be initiated after the Safety Review Committee (SRC) agrees to enter the next dose group based on clinical safety data assessment.

When DLT occurs in 1 of 3 subjects in a dose group, 3 additional subjects in the same dose group will be required (up to 6 subjects in the dose group have completed DLT assessment): if no DLT occurs in the additional 3 subjects, dose escalation will continue; if 1 of the 3 additional subjects experiences one DLT, dose escalation will be discontinued; if more than 1 of the 3 additional subjects experiences DLTs, dose escalation will be discontinued, and 3 additional subjects will be required to be enrolled at one lower dose level for DLT assessment. After the end of escalation for the maximum dose group, if no MTD is observed, the highest dose level is defined as the MTD.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 to 70 years old (inclusive), male or female;
* Expected survival time ≥ 3 months;
* ECOG performance status of 0-1;
* Malignant lymphoma diagnosed according to WHO2016 criteria: priority will be given to T-cell acute lymphoblastic leukemia/lymphoma (including early pre-T-cell lymphoblastic leukemia);
* Subjects with recurrent/refractory T-cell acute lymphoblastic leukemia/lymphoma (including early pre-T-cell lymphoblastic leukemia) who have failed standard treatment or lack effective treatment and meet any of the following criteria:

  1. No remission after at least two courses of standard induction chemotherapy;
  2. Early relapse (<12 months) after complete remission; Or complete remission followed by late relapse (≥12 months) without remission after a course of standard induction chemotherapy;
  3. Patients who did not achieve remission after two or more lines of chemotherapy;
  4. Recurrence after hematopoietic stem cell transplantation.
* Lymphoid hematologic malignancies diagnosed as CD7 positive by flow cytometry and/or CD7 positive by histopathological immunohistochemistry at screening, with the positive rate of tumor ≥ 30%;
* For CD7-positive lymphoid hematologic malignancies involving bone marrow and/or peripheral blood, patients with CD4/CD8 double-negative surface immunophenotype of tumor cells as determined by flow cytometry;
* Liver, kidney and cardiopulmonary function shall meet the following requirements:

  1. Creatinine ≤ 1.5 ULN;
  2. Left ventricular ejection fraction ≥ 45%;
  3. Oxygen saturation > 91%;
  4. Total bilirubin ≤ 2 × ULN; ALT and AST ≤ 2.5 × ULN; for ALT and AST abnormalities due to disease (e.g., liver infiltration or bile duct obstruction) as judged by the investigator, the indicators can be relaxed to ≤ 5 × ULN;
* Patients who can understand the trial and have signed informed consents.

Exclusion Criteria:

* Subjects who need to use immunosuppressants;
* Subjects with malignant tumors other than T-cell hematological malignancies within 5 years prior to screening, with the exception of adequately treated cervical carcinoma in situ, basal cell carcinoma or squamous cell carcinoma, localized prostate cancer after radical surgery, and ductal carcinoma in situ after radical mastectomy;
* Positive for hepatitis B surface antigen (HBsAg) or hepatitis B core antibody (HBcAb) with peripheral blood hepatitis B virus (HBV) DNA titer detection not within the normal reference range; positive for hepatitis C virus (HCV) antibody and peripheral blood hepatitis C virus (HCV) RNA; positive for human immunodeficiency virus (HIV) antibody; positive for cytomegalovirus (CMV) DNA test; positive for syphilis test;
* Severe heart disease: including but not limited to unstable angina, myocardial infarction (within 6 months prior to screening), congestive heart failure (New York Heart Association [NYHA] classification ≥ III), severe arrhythmia;
* Unstable systemic diseases judged by the investigator: including but not limited to serious liver, kidney or metabolic diseases requiring drug treatment;
* Within 7 days prior to screening, there are active or uncontrollable infections requiring systemic therapy (except for mild genitourinary infection and upper respiratory tract infection);
* Pregnant or lactating women, and female subjects who plan to become pregnant within 2 years after cell infusion or male subjects whose partners plan to become pregnant within 2 years after cell infusion;
* Subjects who have received CAR-T therapy or other gene-modified cell therapy prior to screening;
* Subjects who are receiving systemic steroid therapy within 7 days prior to screening or need long-term use of systemic steroid therapy during treatment as judged by the investigator (except for inhalation or topical use);
* Subjects who have participated in other clinical studies within 3 months prior to screening;
* Subjects who have evidence of central nervous system invasion at screening;
* Conditions not eligible for cell preparation as judged by the investigator;
* Other conditions considered unsuitable for enrollment by the investigator.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Estimated)
Dates: Start 2021-12-01 (Actual); Primary Completion 2022-12-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
DLT | About 2 years
  Dose limiting toxicity
MTD | About 2 years
  Maximum tolerated dose

SECONDARY OUTCOMES:
Assessment of the safety after CD7-targeted chimeric antigen receptor T cells infusion (Safety) | About 2 years
  Number of participants with treatment-related adverse events as assessed by CTCAE v5.0.
Assessment of pharmacokinetic (about Cmax) | 28 days
  Assessment of the highest concentration (Cmax) of CD7-targeted chimeric antigen receptor T cells amplified in peripheral blood after administration.
Assessment of pharmacokinetic (about Tmax) | 28 days
  Assessment of the time to reach the highest concentration (Tmax) of CD7-targeted chimeric antigen receptor T cells in peripheral blood after administration.
Assessment of pharmacokinetic (about AUC0-28d) | 28 days
  Assessment of the area under the curve AUC0-28d after administration.
Assessment of pharmacokinetic (about Cmax) | 90 days
  Assessment of the highest concentration (Cmax) of CD7-targeted chimeric antigen receptor T cells amplified in peripheral blood after administration.
Assessment of pharmacokinetic (about Tmax) | 90 days
  Assessment of the time to reach the highest concentration (Tmax) of CD7-targeted chimeric antigen receptor T cells in peripheral blood after administration.
Assessment of pharmacokinetic (about AUC0-90d) | 90 days
  Assessment of the area under the curve AUC0-90d after administration.
PD endpoints | About 2 years
  The proportion and absolute value of CD7-positive cells in peripheral blood at each time point; concentration levels of CAR-T-related serum cytokines such as CRP and IL-6;
To Evaluate Anti-tumour Activity (Overall Survival) | About 2 year
  Defined as the time from start of CD7 CAR-T cell therapy to death (due to any cause);
To Evaluate Anti-tumour Activity (Progression Free Survival) | About 2 year
  Defined as the time from the start of CD7 CAR-T cell therapy to the first disease progression or recurrence or death from any cause.
To Evaluate Anti-tumour Activity (overall response rate) | About 3 months
  Rate of participants who with lymphoma aquire complete response (CR) or partial response (PR) or those who with leukemia CR or CR with incomplete hematologic recovery (CRi).
Immunogenicity endpoints | About 2 years
  Positive rate of human anti-CAR antibody at each time point.
To Evaluate Anti-tumour Activity (duration of response) | About 2 years
  Defined as the time from the first tumor assessment of CR or PR (lymphoma), CR or CRi (leukemia) to the first assessment of disease recurrence or progression or death due to any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Mingzhi Zhang, Doctor, Principal Investigator — The First Affiliated Hospital of Zhengzhou University; Xiaojun Huang, Doctor, Principal Investigator — Peking University People's Hospital; Heng Mei, Doctor, Principal Investigator — Union Hospital, Tongji Medical College, Huazhong University of Science and Technology; Dehui Zou, Doctor, Principal Investigator — Hematology Hospital of Chinese Academy of Medical Sciences (Hematology Research Center of Chinese Academy of Medical Sciences); He Huang, Doctor, Principal Investigator — Zhejiang University
Locations (1):
- PersonGen.Anke Cellular Therapeutice Co., Ltd., Hefei, Anhui, China

IPD SHARING:
Plan to Share IPD: Undecided